CLINICAL TRIAL: NCT00004458
Title: Longitudinal and Biological Study of Childhood Disintegrative Disorder
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Yale University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/13682; YALE-5P01HD0300830; YALE-HIC-5895
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Pervasive Child Development Disorders; Autism
Keywords: autism; childhood disintegrative disorder; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder; Neurologic Manifestations; Mental Disorders; Rare Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
OBJECTIVES:

I. Compare the developmental course (language acquisition, diagnostic stability, predictors of outcome, and restricted interests and behaviors) of childhood disintegrative disorder versus autism and non-autistic developmental delays.

II. Collect data on molecular genetics of proband and family members.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are evaluated with the following questionnaires at ages 2-3 years and again at ages 5-9: The Autism Diagnostic Interview (ADI); The Autism Diagnostic Observation Schedule (ADOS); Assessment of cognitive functioning; Expressive and receptive language; Adaptive functioning; Measures of burden and functional assessment; The Aberrant Behavior Checklist; The Connors Rating Scale - Parent and Teacher version; and Autism Behavior Checklist

An MRI and EEG are performed, and blood samples are collected from patients and family members for molecular genetic studies.

ELIGIBILITY:
* Psychologically diagnosed (DSM-IV) as Childhood Disintegrative Disorder
* No known genetic or medical syndrome (Down syndrome or cerebral palsy)
* Must speak English

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220
Dates: Start 1997-05

CONTACTS AND LOCATIONS:
Overall Officials: Fred Volkmar, Study Chair — Yale University
Locations (2):
- United States (2):
  - Yale Child Study Center, New Haven, Connecticut
  - University of Chicago Cancer Research Center, Chicago, Illinois

REFERENCES:
- [Background] Volkmar FR, Klin A, Marans WD, et al.: Childhood disintegrative disorder. In: Cohen DJ, Volkmar FR.: Handbook of autism and pervasive developmental disorders. 2nd ed., New York, NY: John Wiley, 1997, pp 47-59.